CLINICAL TRIAL: NCT05180435
Title: Family Meals as a Strategy for the Primary Prevention of Cardiovascular Disease in Children
Brief Title: Dietary Approaches for Cardiovascular Health Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1761471
Record Dates: First submitted 2021-12-06; First posted 2022-01-06 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Meals (Experimental): Have at least 5 dinners per week.
  Interventions: Behavioral: Family Meals
- Standard (Active Comparator): Consume the recommended amounts of fruits and vegetables.
  Interventions: Behavioral: Standard

INTERVENTIONS:
Behavioral: Family Meals — A family-based multicomponent lifestyle modification intervention with the goal to increase the frequency of family meals and meet physical activity recommendations.
  Arms: Family Meals
Behavioral: Standard — A family-based multicomponent lifestyle modification intervention with the goal to increase the consumption of fruits and vegetables and and meet physical activity recommendations.
  Arms: Standard

SUMMARY:
The primary purpose of this study is to examine the efficacy of family meal frequency as an intervention target in addressing the primary prevention of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Parents who have a male or female child aged 6-12 years-old with a BMI-for-sex and age <95th percentile
* Parent age is ≥18 years-old
* Parent reports at least 2 of the following CVD risk factors: smoking, high cholesterol, high blood pressure, physical inactivity, overweight/obesity, diabetes
* Parent is able to read, speak and understand English

Exclusion Criteria:

* Parents who live with their child <5 days per week
* Parents who do not have access to the internet and/or are unable to attend intervention sessions
* Parents who report a medical condition that impacts growth or requires a specific eating plan for themselves or their child.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in diet quality. | Baseline and Months 2, 6, 8 and 10
  The Healthy Eating Index is a score ranging from 0-100 with higher scores indicating greater adherence to the Dietary Guidelines.

SECONDARY OUTCOMES:
Change from baseline in body mass index z-scores (zBMI) | Baseline and Months 2, 6, 8 and 10
  Body mass index z-scores (zBMI) will be calculated using Centers for Disease Control and Prevention growth charts. Height will be measured in centimeters and weight will be measured in kilograms and used to calculate BMI as kilograms/meter squared.
Change from baseline in blood pressure | Baseline and Month 6
  Both systolic and diastolic blood pressure.
Change from baseline in fasting insulin | Baseline and Month 6
  Measure of insulin in the blood after fasting.
Change from baseline in fasting glucose | Baseline and Month 6
  Measure of blood sugar (glucose) after fasting.
Change from baseline in lipid levels | Baseline and Month 6
  Nuclear magnetic resonance (NMR) measures of lipoprotein (low-density lipoprotein [LDL], high-density lipoprotein [HDL], very-low density lipoprotein [VLDL]) particle number and size will be assessed.
Change from baseline in pulse wave analysis. | Baseline and Month 6
  PWA will be assessed by a central aortic pressure waveform synthesized from the measured brachial artery pressure waveform via a standard blood pressure cuff inflation/deflation and blood pressure monitoring.
Change from baseline in carotid-to-femoral pulse wave velocity (PVW) | Baseline and Month 6
  Carotid-to-femoral PWV will be measured by simultaneously recording electrocardiography (ECG) and a carotid or femoral pressure waveform via a standard blood pressure cuff inflation/deflation and blood pressure monitoring. The distance from the carotid measurement point to the sternal notch will be subtracted from the distance from the sternal notch to the femoral measurement point and used as propagation distance. PWV will be calculated as propagation distance/time delay. PWV is a measure of regional stiffness of the aorta.
Change in baseline in flow-mediated dilation (FMD) | Baseline and Month 6
  The FMD technique will be employed by assessing the diameter and blood flow velocity of the artery located in the upper arm via ultrasonography. FMD will be used as a measure of endothelial-dependent vessel function and will be expressed as a percent change from baseline, normalized for shear rate calculated from blood flow velocity and vessel diameter data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Energy Balance and Nutrition Laboratory, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No